CLINICAL TRIAL: NCT05949944
Title: Linperlisib in Combination With CHOP in Previously Untreated Peripheral T-Cell Lymphoma：a Single-Arm, Open Lable， Multicenter Clinical Trial（LINCH Study）
Brief Title: Linperlisib in Combination With CHOP in Previously Untreated Peripheral T-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-183
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Linperlisib in combination with CHOP (Experimental): Patients will receive six cycles of induction therapy of linperlisib in combination with CHOP regimen. All patients with CR and PR after induction therapy receive linperlisib maintenance therapy every 28 days until disease progression or other reasons lead to discontinuation, and the duration of linperlisib maintenance does not exceed 24 months.
  Interventions: Drug: Linperlisib in combination with CHOP

INTERVENTIONS:
Drug: Linperlisib in combination with CHOP — Patients will receive six cycles of induction therapy of linperlisib in combination with CHOP regimen. All patients with CR and PR after induction therapy receive linperlisib maintenance therapy every 28 days until disease progression or other reasons lead to discontinuation, and the duration of linperlisib maintenance does not exceed 24 months.

SUMMARY:
This phase Ib/II, single arm, open label, multicenter study is conducted to evaluate the efficacy and safety of linperlisib in combination with CHOP for newly diagnosed PTCL patients, and explore the reasonable dosage of linperlisib when combined with CHOP regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed PTCL, including peripheral T-cell lymphoma non-specific type (PTCL NOS), angioimmunoblastic T-cell lymphoma (AITL), enteropathy related T-cell lymphoma and liver spleen T-cell lymphoma;
2. Has not received anti-tumor treatment in the past;
3. There must be at least one evaluable lesion/measurable lesion according to the 2014 Lugano Lymphoma Evaluation Criteria. An evaluable lesion is defined as a lymph node or extra-nodal local lesion that shows increased uptake of 18FDG on PET-CT (higher than the liver), with lesion characteristics consistent with lymphoma manifestations. A measurable lesion is defined as a nodule with a longest diameter of >15mm or an extra-nodal lesion with a longest diameter of >10mm, accompanied by increased uptake of 18FDG. Exclusion of cases without measurable lesions and diffuse uptake of 18FDG in the liver is required;
4. Age ≥18 years old, regardless of gender;
5. Whole body physical condition score (ECOG) 0-2;
6. Expected survival time>3 months;
7. Adequate bone marrow and organ functions;
8. Not accompanied by hemophagocytic syndrome; If the patient is accompanied by clinically diagnosed hemophagocytic syndrome, after targeted anti hemophagocytic syndrome drug treatment, the researcher evaluates the patient's general physical condition to determine whether they can be enrolled.
9. Volunteer to participate in clinical research and sign an informed consent form, willing to follow and capable of completing all trial procedures.

Exclusion Criteria:

1. Received PI3K inhibitor treatment before enrollment;
2. A history of other primary invasive malignant tumors that have not been relieved or have not been relieved for more than 3 years;
3. Involvement of the central nervous system (meninges or brain parenchyma);
4. Individuals who are known to have allergies to any medication in the study
5. Participated in clinical trials of other drugs within 4 weeks prior to the start of the study;
6. Pregnant or lactating women;
7. Individuals with active infections, excluding fever related to tumor B symptoms;
8. Concomitant diseases and medical history:

   1. There are many factors affecting oral medicine (such as inability to swallow, chronic diarrhea and Bowel obstruction);
   2. Individuals with a history of abuse of psychotropic substances who are unable to quit or have mental disorders;
   3. Subjects with any severe and/or uncontrollable diseases, including:

      1. Poor blood pressure control (systolic blood pressure ≥ 150mm Hg or diastolic blood pressure ≥ 100 mmHg);
      2. Suffering from ≥ Level 2 myocardial ischemia or infarction, arrhythmia (including QTc ≥ 450ms (male), QTc ≥ 470ms (female)), and ≥ Level 2 congestive heart failure (New York Heart Association (NYHA) classification);
      3. Active interstitial pneumonia or other chronic lung diseases, leading to severe impairment of lung function, defined as FEV1 and DLCOc<60% of normal predicted values; A history of interstitial pneumonia caused by COVID-19.
      4. Liver abnormalities:

         I. Decompensated cirrhosis (Child Pugh liver function rating of B or C) II Known clinically significant history of liver disease. Including viral hepatitis, known carriers of hepatitis B virus (HBV) must exclude active HBV infection, i.e. HBV DNA positivity (>2500 copies/mL or>500IU/mL, and greater than the upper limit of normal values); Known hepatitis C virus infection (HCV) and HCV RNA positivity (>1 × 103 copies/mL). Note: hepatitis B HBsAg positive subjects who meet the inclusion conditions, whether their HBV DNA is measurable or not, need to continue antiviral treatment (nucleoside analogues are recommended) and regularly monitor HBV DNA; For subjects with positive HBcAb but negative HBsAg in hepatitis B, HBV DNA should be monitored regularly and preventive antiviral treatment should be recommended; Hepatitis C patients need to regularly monitor HCV RNA.
      5. Renal failure requiring hemodialysis or Peritoneal dialysis;
      6. Subjects with uncontrolled Pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
      7. Poor control of diabetes (Fasting blood sugar (FBG)>10mmol/L);
      8. Urinary routine examination indicates that urine protein is ≥++, and it is confirmed that 24-hour urine protein quantification is greater than 1.0 g;
9. . Have a history of immune deficiency, including positive Diagnosis of HIV/AIDS, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation;
10. . According to the judgment of the researcher, there are serious accompanying diseases that pose a serious threat to the patient's safety or affect the patient's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT, Phase Ib) | The first cycle of linperlisib in combination with R-CHOP regimen (21 days)
  To identify the DLT
Complete remission rate (CR rate) based on the 2014 Lugano evaluation criteria (Phase II) | Up to 18 weeks
  To investigate the antitumor efficacy

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 18 weeks
  To investigate the antitumor efficacy
Duration of complete remission | From date of complete remission to the study treatment until the date of the first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To investigate the antitumor efficacy
Duration of remission (DOR) | From date of remission to the study treatment until the date of the first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To investigate the antitumor efficacy
Progression free survival (PFS) | From date of the first injection until the date of the first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To investigate the antitumor efficacy
Overall survival (OS) | From date of the first injection until the date of death from ant cause, assessed up to 24 months
  To investigate the antitumor efficacy
Incidence and severity of adverse events (AE) and Serious adverse event (SAE), as well as abnormal laboratory inspection indicators; Quality of Life (QOL). | Through study completion, an average of 2 years
  To identify the incidence of AE, SAE and QOL.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University, Guangzhou, Guangdong, China